CLINICAL TRIAL: NCT04735549
Title: Correction of Vulvovaginal Atrophy in Postmenopausal Women Using Neodymium Laser Treatment
Brief Title: Vulvovaginal Atrophy Correction Using Neodymium Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MeLSyTech, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VACUNL-2020
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal Period; Vaginal Atrophy; Female Urogenital Diseases
Keywords: Vaginal Atrophy; Female Urogenital Diseases; Neodymium Laser; Laser Treatment; Nanosecond; Laser; Vaginal; Postmenopausal
MeSH Terms: conditions — Female Urogenital Diseases | interventions — Laser Therapy; Vaginal Smears; Elasticity Imaging Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The treatment method cannot be hidden from the participants and the researcher because of the very different method of treatment: laser treatment and the use of local hormones on their own. However, the specialists involved in the study (cytologist and ultrasound specialist) will not know which group the participant belongs to. The researcher will refer participants (or their materials) to these specialists, indicating their name and visit number. The Researcher will keep a document matching the participant's name and number.
  The conversation will be held with participants. A participant must not disclose his group when visiting an ultrasound specialist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Treatment (Experimental): Laser treatment of the vagina, vulva, and paraurethral region with a "Magic Max" laser ("Magic Gyno"). In total, three procedures will be performed with an interval of 4-6 weeks.
  During the procedure, the following sequence of actions will be performed: 1st Stage - vaginal processing with a conical mirror handpiece, 2nd Stage - vaginal processing with a corner mirror handpiece, 3d Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.
  Interventions: Device: Laser Treatment; Diagnostic Test: Сlinical blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Vaginal smear; Diagnostic Test: Pelvic ultrasound; Other: Female Sexual Function Index; Other: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire; Other: Vulvovaginal Symptoms Questionnaire; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Elastography (ultrasound investigation); Diagnostic Test: Perineometry; Other: Visual Analogue Scale (VAS)
- Topical hormone (Active Comparator): Local hormone therapy with estriol. The course of treatment will be of 2 weeks of daily use, and then a maintenance therapy for 12 months to prevent symptoms.
  Interventions: Drug: Topical hormone estriol; Diagnostic Test: Сlinical blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Vaginal smear; Diagnostic Test: Pelvic ultrasound; Other: Female Sexual Function Index; Other: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire; Other: Vulvovaginal Symptoms Questionnaire; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Elastography (ultrasound investigation); Diagnostic Test: Perineometry; Other: Visual Analogue Scale (VAS)
- Laser Treatment + Topical hormone (Experimental): Laser treatment of the vagina, vulva, and paraurethral region with a "Magic Max" laser ("Magic Gyno"). In total, three procedures will be performed with an interval of 4-6 weeks. During the procedure, the following sequence of actions will be performed: 1st Stage - vaginal processing with a conical mirror handpiece, 2nd Stage - vaginal processing with a corner mirror handpiece, 3d Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.
  At the same time local hormone therapy with estriol. The course of treatment will be of 2 weeks of daily use, and then a maintenance therapy for 12 months to prevent symptoms.
  Interventions: Device: Laser Treatment; Drug: Topical hormone estriol; Diagnostic Test: Сlinical blood analysis; Diagnostic Test: Сlinical urine test; Diagnostic Test: Vaginal smear; Diagnostic Test: Pelvic ultrasound; Other: Female Sexual Function Index; Other: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire; Other: Vulvovaginal Symptoms Questionnaire; Diagnostic Test: Vaginal Health Index; Diagnostic Test: Elastography (ultrasound investigation); Diagnostic Test: Perineometry; Other: Visual Analogue Scale (VAS)

INTERVENTIONS:
Device: Laser Treatment — Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 ns, the pause between pulses is 30 us. The energy of one pulse is about 1 mJ.
  General laser radiation parameters for 1st and 2nd stages are: beam with diameter of 4 millimeters (mm) scans treatment area by 4 circles with step of 2 mm (50 percentage (%) overlap), average power of 10-25 Watt (W), treatment time in one point of 1-10 seconds (s), treatment step of 5 mm, from 1 to 5 repetitions of total vagina treatment. General laser radiation parameters for 3d stage are: beam diameter of 6 mm, average power of 15-30 W, duration of ns-pulses packet of 50-100 milliseconds (ms), pause between packets of 50-100 ms, treatment duration up to 65 s, treatment in permanent motion with speed of 10-50 mm/s.
  The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.
  Arms: Laser Treatment; Laser Treatment + Topical hormone
Drug: Topical hormone estriol — Estriol ((17 beta)-estra-1,3,5 (10)-trien-3,17-diol). Daily dose will be 0.5 gram daily for 2 weeks, later 0.5 gram twice a week for 12 months.
  Arms: Laser Treatment + Topical hormone; Topical hormone
Diagnostic Test: Сlinical blood analysis — Taking blood from a vein for Clinical blood analysis, Wassermann reaction (WR), human immunodeficiency viruses (HIV), hepatitis B infection (HBsAg), hepatitis C infection (HCVAg) determination, glucose test (to include the participant in the study).
Diagnostic Test: Сlinical urine test — Urine sampling for Clinical urine test (to include the participant in the study).
Diagnostic Test: Vaginal smear — Vaginal smear for flora investigation (to include the participant in the study), cytology, microbiological analysis with Gram staining (to evaluate procedure efficiency).
Diagnostic Test: Pelvic ultrasound — Pelvic ultrasound investigation to determine pathologies of the pelvic through a gynecological probe (to include the participant in the study).
Other: Female Sexual Function Index — Female Sexual Function Index will be used to collect feedback on changes in the participants life quality (to evaluate procedure efficiency).
Other: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire — The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire will be used to collect feedback on changes in the participants life quality (to evaluate procedure efficiency).
Other: Vulvovaginal Symptoms Questionnaire — Vulvovaginal Symptoms Questionnaire will be used to collect feedback on changes in the participants life quality (to evaluate procedure efficiency).
Diagnostic Test: Vaginal Health Index — Vaginal Health Index will be investigated by clinical examination for vaginal elasticity, vaginal secretions, epithelial mucous membrane, vaginal hydration. Potential of hydrogen (pH) will be investigated by test-lines paper (to evaluate procedure efficiency).
Diagnostic Test: Elastography (ultrasound investigation) — Ultrasound investigation for assessing elasticity / stiffness of tissues of vulva region with Mindray device (head L14-6WU) (to evaluate procedure efficiency).
Diagnostic Test: Perineometry — Pressure force of vaginal walls measurement with EmbaGYN device (to evaluate procedure efficiency).
Other: Visual Analogue Scale (VAS) — Visual Analogue Scale will be used to collect feedback on changes in the participants life quality (to evaluate procedure efficiency).

SUMMARY:
The aim of this prospective study is characteristic of changes in the vaginal wall and vulva after treatment of neodymium laser radiation with a wavelength of 1064 nm. To assess the condition of the vaginal walls and vulva before and after laser treatment, the following methods will be used: vaginal health index, perineometry, elastography of vulva, cytological methods. Female Sexual Function Index (FSFI), The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12), Vulvovaginal Symptoms Questionnaire (VSQ), Visual Analogue Scale (VAS) will be used to collect feedback on changes in the participants life quality. Total up to 120 participants with postmenopausal atrophy will be involved in the study. Participants will be divided into three groups: laser treatment group, topical hormones treatment group, and both laser treatment with topical hormones application group, by 40 participants in each. The time intervals between tests will be the same for all groups. Thus, a direct comparison between conventional treatment (topical hormones), laser treatment and combine laser and topical hormones therapy of the vaginal atrophy will be made. The main hypothesis of the study is improvement in condition of the vaginal walls after laser treatment and laser treatment with hormones application compared with the initial state of not less than thirty percent of participants, and improvement in condition on average compared with the hormones only therapy group.

DETAILED DESCRIPTION:
The principle of participant distribution into groups is the main method of treatment of postmenopausal vaginal atrophy. Total up to 120 participants with postmenopausal atrophy will be involved in the study. Participants will be divided into three groups: laser treatment group, topical hormones treatment group, laser treatment with topical hormones application, by 40 participants in each.

The types of examination of each group are the same and include:

General methods: physical examination, clinical blood analysis with glucose determination, clinical urine test, vaginal smear for flora and oncocytology, pelvic ultrasound.

Special methods: filling out the questionnaire (Female Sexual Function Index, The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, Vulvovaginal Symptoms Questionnaire), Vaginal Health Index determination, Visual Analogue Scale (VAS) determination, perineometry, vaginal smear for cytology, elastography of vulva, microbiological vaginal smear stained by Gram.

The treatment procedure of this study is the laser treatment of the vagina and vulva with a "Magic Max" laser ("Magic Gyno" from August 2024) with subsequent monitoring.

Treatment Technique:

Laser treatment procedure will be carried out in three stages. In total, three procedures will be performed with an interval of 4-6 weeks. Two follow-up visits will follow: 1 and 6 months after the last procedure.

During the procedure, the following sequence of actions will be performed:

1. st Stage - vaginal processing with a conical mirror handpiece,
2. nd Stage - vaginal processing with a corner mirror handpiece,
3. rd Stage - external vulva and paraurethral region processing with a switched beam diameter handpiece.

Laser radiation is emitted by a series of pulses following each other through a pause. The duration of one pulse is 20-200 nanoseconds (ns), the pause between pulses is 30 microseconds (us). The energy of one pulse is about 1 millijoule (mJ). The procedure is performed without anesthesia. The doctor always focuses on the participant's feeling of warmth.

Hormone treatment procedure. Local hormone therapy with estriol will be used as a therapeutic tool for the control group. The course of treatment will be of 2 weeks of daily use, and then a maintenance therapy will be used of 2 times a week for 12 months to prevent symptoms.

Participants of all groups will be tested with the general methods necessary to include the participant in the study at the first visit.

For the laser treatment group: Studies will be carried out using special methods and then laser treatment of the vagina and vulva and paraurethral region will be performed during the 2nd, 3d, and 4th visits. Studies with all special methods will be performed during the 1st (before the start of treatment) visit. Vaginal health index, pH-measurement, perineometry, and filling of questionnaires will be performed during 3d-6th visits. Cytological investigation and elastography of vulva will be performed during 5th (1 month after the last procedure) and 6th (6 months after the last procedure).

For the hormone treatment group: Studies with all special methods will be performed during the 1st (before the start of treatment) visit. Vaginal health index, pH-measurement, perineometry, and filling of questionnaires will be performed during 3d-6th visits. Cytological investigation and Doppler sonography will be performed during 5th (1 month after the last procedure) and 6th (6 months after the last procedure). Hormone therapy will begin from the 2nd visit. All subsequent visits will be carried out at the same time intervals as for the laser treatment group, using studies with special methods. The 3d visit will be in 4-6 weeks after the start of treatment, the 4th will be in 4-6 weeks after the 3d visit, the 5th - 1 month after the 4th, the 6th - 6 months after the 4th.

For the combine laser treatment with topical hormones application group: laser treatment of the vagina and vulva and paraurethral region will be performed during the 2nd, 3d, and 4th visits. At the same time, starting from 2nd visit hormone therapy will be started. All subsequent visits will be carried out at the same time intervals as for the laser treatment group and hormone treatment group, using studies with special methods.

Thus, a direct comparison between conventional treatment (topical hormones), laser treatment and combine therapy of the vaginal atrophy will be made during the treatment, as well as on follow-up visits in 1 and 6 months after the end of each type of treatment.

The study will be carried out with the participation of FSBI "National Medical Research Center For Obstetrics, Gynecology And Perinatology Named After Academician V.I.Kulakov" MINISTRY OF HEALTHCARE OF THE RUSSIAN FEDERATION

All data obtained during the study will be transferred to the manufacturer of "MeLSyTech" Ltd.

The study will be monitored by "MeLSyTech" Ltd as follows:

* Once a month, monitoring of provided documents (copies of individual registration records of participants, informed consent, test results) for the complete filling of the forms; the clarity of filling out forms, the possibility of systematizing information from the forms of their assessment;
* Once every six months, monitoring will be conducted with a coordinator visit of the research center and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management;
* Once a year, the investigator submits a clinical evaluation report to the sponsor.

Statistics

The analysis will be carried out both between groups of participants receiving different types of therapy (analysis of independent groups) and within groups at different time intervals (analysis of matched groups).

Before performing statistical analysis of the data, the distribution type of the variables will be assessed. To assess the normality of distribution for each variable, histograms of frequency distributions will be visually evaluated, indicators of skewness, kurtosis, and the D'Agostino-Pearson normality test will be used.

In addition to checking the type of distribution of variables, the equality of variances of the studied groups will be assessed using the methods of analysis of variance, in particular the Brown-Forsythe test.

Methods of descriptive analysis will be used depending on the type of distribution of the variable. With a normal distribution, the mean (M) and standard deviation (SD) will be calculated. In case of an nongaussian distribution, the median (Me) and interquartile range will be calculated. Different algorithms of statistical analysis will be applied depending on the type of distribution of variables.

Comparison of the paired and unpaired groups with a normal distribution, in case of the equality of the variances, will be carried out by the methods of analysis of variance ANOVA. Comparison of groups in pairs will be performed using the post-hoc method of posterior multiple comparisons (Tukey test).

Comparison of groups in which variables do not follow the normal distribution will be carried out using the methods of nonparametric analysis of variations: the Kruskal-Wallis test (ANOVA tests) for independent groups and the Friedman test for matched groups. Dunn's multiple comparison test will be used to assess intergroup differences.

Before assessing intergroup differences, the initial samples (1 visit) will be analyzed for identity using ANOVA or nonparametric Kruskal-Wallis tests (depending on the type of data). In case of significant differences in the samples, the search and removal of extremely deviating values (outliers) will be carried out.

Differences will be considered statistically significant if the significance P values are <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age of over 50 years old, inclusive;
* Participants diagnosed with genitourinary menopausal syndrome with severe signs of vulvovaginal atrophy;
* Participants were examined according to the proposed protocol;
* Participants who signed informed consent and fully informed about the purpose of the study.

Exclusion Criteria:

* Tendency to photoallergy including taking photosensitizing drugs (diuretics, antihistamines, antipsychotics);
* Porphyria;
* Active tuberculosis;
* Damage to the vaginal mucosa;
* Urinary tract infections in the acute stage;
* Genital herpes in the acute stage;
* Inflammatory diseases of the vulva and vagina in the acute stage;
* Oncological diseases of the female reproductive system, including history of oncological diseases;
* Precancerous diseases of the cervix, vagina and vulva;
* The use of drugs and other methods of treatment (including laser) that can affect the result, less than 1 month before the start of the study and during the study (Menopausal hormone therapy, the use of topical estriol; Kegel exercises, physiotherapy, the use of pelvic floor muscle trainers).
* Protocol non-compliance of laser exposure sessions;
* Voluntary refusal to participate in the study;
* Violation of recommendations for the management of the period after laser treatment;
* Adverse events that occurred during laser processing and research, and associated with them.
* The occurrence of adverse events or other symptoms that are contraindications to laser procedures, as well as the occurrence of cases described in the exclusion criteria.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline of Vaginal Health Index Score | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Vaginal Health Index will be investigated by clinical examination for vagina:
  A. Vaginal elasticity (Characteristic=Points: Non=1, Poor=2, Fair=3, Good=4, Excellent=5), B. Vaginal secretions (None=1; Sсant, thin yellow=2; Superficial, thin white=3; Moderate, thin white=4; Normal (white)=5), C. Epithelial mucous membrane (Petechiae noted before contact=1, Bleeding with light contact=2, Bleeds with scraping, Not friable thin epithelium=4, Normal=5), D. Vaginal hydration (None, surface inflamed=1, None, surface nod inflamed=2, Minimal=3, Moderate=4, Normal=5), E. pH will be investigated by test-lines paper (≥6.1=1, 5.6-6.0=2, 5.1-5.5=3, 4.7-5.0=4, ≤4.6=5).
  Score=A+B+C+D+E

OTHER OUTCOMES:
Mean Change from Baseline of "Desire" Score on the Female Sexual Function Index Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Participants answer questions:
  Q1. Over the past 4 weeks, how often did you feel sexual desire or interest? Answers = Points: almost always or always (5), most times (more than half the time) (4), sometimes (about half the time) (3), a few times (less than half the time) (2), almost never or never (1).
  Q2. Over the past 4 weeks, how would you rate your level (degree) of sexual desire or interest? Answers = Points: very high (5), high (4), moderate (3), low (2), very low or none at all (1)
  Score = (Score to Q1 + Score to Q2)*0.6
Mean Change from Baseline of "Arousal" Score on the Female Sexual Function Index Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Participants answer questions: Q3. Over the past 4 weeks, how often did you feel sexually aroused during sexual activity or intercourse? Q6. Over the past 4 weeks, how often have you been satisfied with your arousal (excitement) during sexual activity or intercourse? Answers = Points (Q3 and Q6): no sexual activity (0), almost always or always (5), most times (4), sometimes (3), a few times (2), almost never or never (1) Q4. Over the past 4 weeks, how would you rate your level of sexual arousal during sexual activity or intercourse? Answers = Points: no sexual activity (0), very high (5), high (4), moderate (3), low (2), very low or none at all (1) Q5. Over the past 4 weeks, how confident were you about becoming sexually aroused during sexual activity or intercourse? Answers=Points: no sexual activity (0), very high confidence (5), high confidence (4), moderate confidence (3), low confidence (2), very low or no confidence (1) Score=(Score to Q3+Score to Q4+Score to Q5+Score to Q6)*0.3
Mean Change from Baseline of "Lubrication" Score on the Female Sexual Function Index Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Participants answer questions:Q7. Over the past 4 weeks, how often did you become lubricated ("wet") during sexual activity or intercourse?Q9. Over the past 4 weeks, how often did you maintain your lubrication ("wetness") until completion of sexual activity or intercourse?Answers = Points: no sexual activity (0), almost always or always (5), most times (more than half the time) (4), sometimes (about half the time) (3), a few times (less than half the time) (2), almost never or never (1). Q8. Over the past 4 weeks, how difficult was it to become lubricated ("wet") during sexual activity or intercourse? Q10. Over the past 4 weeks, how difficult was it to maintain your lubrication ("wetness") until completion of sexual activity or intercourse? Answers = Points: no sexual activity (0), extremely difficult or impossible (1), very difficult (2), difficult (3), slightly difficult (4), not difficult (5). Score = (Score to Q7 + Score to Q8 + Score to Q9 + Score to Q10)*0.3
Mean Change from Baseline of "Orgasm" Score on the Female Sexual Function Index Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Participants answer questions:
  Q11. Over the past 4 weeks, when you had sexual stimulation or intercourse, how often did you reach orgasm (climax)? Answers = Points: no sexual activity (0), almost always or always (5), most times (4), sometimes (3), a few times (2), almost never or never (1).
  Q12. Over the past 4 weeks, when you had sexual stimulation or intercourse, how difficult was it for you to reach orgasm (climax)? Answers = Points: no sexual activity (0), extremely difficult or impossible (1), very difficult (2), difficult (3), slightly difficult (4), not difficult (5).
  Q13. Over the past 4 weeks, how satisfied were you with your ability to reach orgasm (climax) during sexual activity or intercourse? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Score = (Score to Q11 + Score to Q12 + Score to Q13)*0.4
Mean Change from Baseline of "Satisfaction" Score on the Female Sexual Function Index Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Participants answer questions:
  Q14. Over the past 4 weeks, how satisfied have you been with the amount of emotional closeness during sexual activity between you and your partner? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Q15. Over the past 4 weeks, how satisfied have you been with your sexual relationship with your partner? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Q16. Over the past 4 weeks, how satisfied have you been with your overall sexual life? Answers = Points: no sexual activity (0), very satisfied (5), moderately satisfied (4), about equally satisfied and dissatisfied (3), moderately dissatisfied (2), very dissatisfied (1).
  Score = (Score to Q14 + Score to Q15 + Score to Q16)*0.4
Mean Change from Baseline of "Pain" Score on the Female Sexual Function Index Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Participants answer questions:
  Q17. Over the past 4 weeks, how often did you experience discomfort or pain during vaginal penetration? Answers = Points: did not attempt intercourse (0), almost always or always (1), most times (2), sometimes (3), a few times (4), almost never or never (5).
  Q18. Over the past 4 weeks, how often did you experience discomfort or pain following vaginal penetration? Answers = Points: did not attempt intercourse (0), almost always or always (1), most times (2), sometimes (3), a few times (4), almost never or never (5).
  Q19. Over the past 4 weeks, how would you rate your level (degree) of discomfort or pain during or following vaginal penetration? Answers = Points: did not attempt intercourse (0)very high (1)high (2)moderate (3)low (4)very low or none at all (5).
  Score = (Score to Q17 + Score to Q18 + Score to Q19)*0.4
Mean Change from Baseline of "Sexual Function in Women with Urinary Incontinence and/or Pelvic Organ Prolapse" Score on Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Q1 How frequently do you feel sexual desire?Q2 Do you climax when having sexual intercourse with your partner?Q3 Do you feel sexually excited when having sexual activity with your partner?Q4 How satisfied are you with the variety of sexual activities in your sex life?Q5 Do you feel pain during sexual intercourse?Q6 Are you incontinent with sexual activity?Q7 Does fear of incontinence restrict your sexual activity?Q8 Do you avoid sexual intercourse because of bulging in the vagina?Q9 When you have sex with your partner, do you have negative emotional reactions such as fear, disgust, shame or guilt?Q10 Does your partner have a problem with erections that affects your sexual activity?Q11 Does your partner have a problem with premature ejaculation that affects your sexual activity?Q12 Compared to orgasms you have had in the past, how intense are the orgasms you have had in the past six months?Answers=never(4),seldom(3),sometimes(2),usually(1),always(0).Inverted scale for questions 1-4
Mean Change from Baseline of "Disease-Specific Quality-of-Life Impact of Vulvovaginal Symptoms in Postmenopausal Women" Score on The Vulvovaginal Symptom Questionnaire | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Participants answer questions:
  Q1. Your vulva itching? Q2. Your vulva burning or stinging? Q3. Your vulva hurting? Q4. Your vulva being irritated? Q5. Your vulva being dry? Q6. Discharge from your vulva or vagina? Q7. Odor from your vulva or vagina? Q8. Worry about your vulvar symptoms (VS)? Q9. The appearance of your vulva? Q10. Frustration about your VS? Q11. Embarrassment about your VS? Q12. The effects of your VS on your interactions with others? Q13. The effects of your VS on your desire to be with people? Q14. Your VS making it hard to show affection? Q15. The effects of your VS on your daily activities? Q16. Your VS affecting your desire to be intimate? Q17. Are you currently sexually active with a partner? Q18. The effects of your VS on your sexual relationships? Q19. Your VS causing pain during sexual activity? Q20. Your VS causing dryness during sexual activity? Q21. Your VS causing bleeding during sexual activity?
  Answers = Points: no (0), yes (1)
Mean Change from Baseline of Compression Time of Vagina | [Time Frame: 1st visit (before any treatment); 2nd visit (first treatment) 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Measurement is a part of perineometry. Participants will be asked to hold the EmbaGYN device bulb with maximum pressure they can. Compression Time will be measured with EmbaGYN device as inner function, in seconds (s).
Mean Change from Baseline of Maximum Pressure at Contraction of Vagina | [Time Frame: 1st visit (before any treatment); 2nd visit (first treatment) 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Measurement is a part of perineometry. Participants will be asked to hold the EmbaGYN device bulb with maximum pressure they can. Maximum pressure at contraction will be measured with EmbaGYN device as inner function, in millimeter of mercury column (mmHg).
Mean Change from Baseline of Average Pressure at Contraction of Vagina | [Time Frame: 1st visit (before any treatment); 2nd visit (first treatment) 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Measurement is a part of perineometry. Participants will be asked to hold the EmbaGYN device bulb with maximum pressure they can. Average pressure at contraction will be measured with EmbaGYN device as inner function, in millimeter of mercury column (mmHg).
Mean Change from Baseline of Maturation Index in vaginal smear | [Time Frame: 1st visit (before any treatment); 1 month after 4th visit and 6 months after 4th visit]
  Part of a cytological test. Prior to coding the Maturation Index (MV), the coder counts 100 cells in aliquot and records the proportion of parabasal (P), intermediate (I), and superficial (S) cells. The Maturation Index are calculated using formula: the percentage of superficial cells (S) plus 0.5 times the percentage of intermediate cells (I) coded from the cytology sample [MV= %S + (0.5 × % I)].
Mean Change from Baseline of Stiffness of Tissues of Vulva | [Time Frame: 1st visit (before any treatment); 1 month after 4th visit and 6 months after 4th visit]
  Elastography wirh ultrasound investigation. The stiffness of soft tissues will be measured in 4 points: in the area of the middle of the connection of the labia majora and labia minora on both sides and in the area of the middle of the inner surface of the labia minora on both sides.
  Investigation will be handled with using of ultrasound device Mindray with head L14-6WU. Measure units - kiloPascal (kPa).
Mean Change from Baseline of Visual Analogue Scale score | [Time Frame: 1st visit (before any treatment); 3d visit (4-6 weeks after 2nd visit); 4th visit (4-6 weeks after 3d visit) - the end of laser treatment; 1 month after 4th visit and 6 months after 4th visit]
  Q1.1 Burning in the vulva? Q1.2 Burning in the vagina? Q2.1 Pain in the vulva? Q2.2 Pain in the vagina? Q3.1 Itching in the vulva? Q3.2 Itching in the vagina? Q4.1 Dryness in the vulva? Q4.2 Dryness in the vagina? Q5.1 Pain in the vulva during sexual activity? Q5.2 Pain in the vagina during sexual activity? Q6 Frequent urge to urinate? Q7 Urinary incontinence with an imperative urge to urinate? Q8 Urinary incontinence when coughing/sneezing/lifting heavy/exercise, etc.? Answers = Visual Analogue Scale, where No (0), Always bother (10). Total Score = SUM(Q1.1-Q8)
Mean Change from Baseline of Vaginal Smear Microbiologic investigation with Gram staining score. | [Time Frame: 1st visit (before any treatment); 1 month after 4th visit and 6 months after 4th visit]
  Smear will be sampled from the posterior wall of vagina and stained according to Gram. For estimation of grade of bacterial vaginosis criteria or the Nugent will be used. Morphotypes of Lactobacilli, Gardnerella and Mobiluncus in swear will be counted. General score will be counted by following equation:
  A (Lactobacilli morphotypes) = 0(>30), 1(5-30), 2(1-4), 3(1), 4(0) B (Gardnerella morphotypes) = 0(0), 1(1), 2(1-4), 3(5-30), 4(>30) C (Mobiluncus morphotypes) = 0(0), 1(1), 2(1-4), 3(5-30), 4(>30) General score = A+B+C

CONTACTS AND LOCATIONS:
Overall Officials: Inna A Apolikhina, Ph.D., Principal Investigator — Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov
Locations (1):
- Federal State Budget Institution "National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov", Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
The following data can be shared with researchers upon an official request:
  The final version of the Study Protocol approved by the Local Ethics Committee; Copies of anonymized filled Individual Registration Cards (IRC); Informed Consent Form (ICF); Clinical Study Report (CSR) and/or published article (if not contradict the rules and conditions of a journal); Supplement files systematizing data.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD can be shared with researchers starting 3 months after CSR or article publication for five years.
Access Criteria: IPD can be shared with researchers only upon an official request from researcher's affiliation institution in the letter form on organization's letterhead paper signed by an authorized person. Official request must be directed by e-mail to the contact person (Ksenia Shatilova, shatilova@melsytech.com). The letter must contain the request purpose and statement of internal IPD use as confidential information only.
  IPD will be shared after approval by CEO of "MeLSyTech" Ltd according to the company internal rules. A requester will be notified of the decision by official letter. Depending on the decision, a requester will receive a link to the repository, or a justified rejection.